CLINICAL TRIAL: NCT06445517
Title: A Phase 1, Open-label, Multicenter, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of ISM8207 Monotherapy in Patients With Advanced Solid Tumors or Relapsed/Refractory B-Lymphoid Malignancies
Brief Title: Study Evaluating ISM8207 in Participants With Advanced Solid Tumors and Relapsed/Refractory B-Cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: InSilico Medicine Hong Kong Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ISM8207_101
Record Dates: First submitted 2024-05-31; First posted 2024-06-06 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumors; Relapsed/Refractory B-cell Lymphoma
Keywords: Advanced solid tumors; Relapsed/refractory B-cell lymphoma; Lymphoma, B-cell
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation: ISM8207 (Experimental): Participants will receive ISM8207 orally once on day 1 during single dose period (3 days) then once daily in repeated 28-day cycles from Cycle 1 onwards.
  Interventions: Drug: ISM8207
- Dose Expansion: ISM8207 (Experimental): Participants will receive ISM8207 orally once daily in repeated 28-day cycles.
  Interventions: Drug: ISM8207

INTERVENTIONS:
Drug: ISM8207 — Pharmaceutical formulation: Capsules Mode of Administration: Oral

SUMMARY:
The goal of this clinical trial is to study ISM8207 in participants with advanced solid tumors and relapsed/refractory B-cell lymphoma. The primary objective is to evaluate the safety and tolerability of ISM8207 orally administered in participants with advanced solid tumors and relapsed/refractory B-cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants with age ≥18 years at the time of signing the informed consent.
2. Advanced solid tumors: Histologically confirmed advanced or metastatic solid tumors who have disease progression after standard therapy, intolerable to standard therapy, or for whom no standard therapy exists.

   B-cell lymphoma: Histologically confirmed B-cell lymphoma who had received at least one prior line of standard therapy and were relapsed after or refractory to the standard therapy.
3. Have measurable or evaluable lesions in Part 1 and at least one measurable target lesion in Part 2 as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria or Lugano 2014.
4. ECOG PS (Eastern Cooperative Oncology Group Performance Status)≤1.
5. Life expectancy of ≥12 weeks as judged by the investigator.
6. Adequate organ function as determined by medical assessment.
7. Capable of providing signed ICF and complying with the requirements and restrictions listed in the ICF and in this study protocol.
8. Female subjects of childbearing potential and male subjects must agree to use an effective method of contraception during the treatment period and for 90 days after the last dose of ISM8207.

Exclusion Criteria:

1. Prior treated with other QPCTL, CD47 or SIRPα inhibitors.
2. Burkitt lymphoma/leukemia, plasma cell myeloma, plasmablastic lymphoma.
3. Participation in other therapeutic clinical studies within 28 days or 5 half- lives (whichever is shorter) prior to first dose of study treatment.
4. Anti-tumor therapy (chemotherapy, immunotherapy, targeted therapy, biologic therapy, or other anti-tumor therapy) within 28 days or 5 half-lives, whichever is shorter prior to first dose of study treatment.
5. Previous allogeneic stem cell transplantation or autologous stem cell. transplantation within 3 months prior to first receiving study treatment.
6. Unresolved toxicity of Grade >1 attributed to any prior therapies (excluding alopecia).
7. Received antitumor steroid therapy within 7 days prior to the first study treatment administration.
8. A serious illness or medical condition(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) events | 31 days
Incidence and severity of adverse events (AEs) | Approximately 2 years
Recommended phase 2 dose (RP2D) | 31 days

SECONDARY OUTCOMES:
objective response rate (ORR) | Approximately 2 years
best objective response (BOR) | Approximately 2 years
duration of response (DoR) | Approximately 2 years
disease control rate (DCR) | Approximately 2 years
progression-free survival (PFS) | Approximately 2 years
6-month overall survival (OS) rates | Approximately 2 years
1-year overall survival (OS) rates | Approximately 2 years
maximum observed concentration (Cmax) | Approximately 2 years
time of maximum observed concentration (Tmax) | Approximately 2 years
area under the concentration-time curve (AUC) | Approximately 2 years
terminal half-life (t1/2) | Approximately 2 years
apparent clearance (CL/F) | Approximately 2 years
apparent volume of distribution (Vz/F) | Approximately 2 years
maximum observed concentration at steady state (Css,max) | Approximately 2 years
minimum observed concentration at steady state (Css,min) | Approximately 2 years
average concentration at steady state (Css,av) | Approximately 2 years
time of Css,max (Tss,max) | Approximately 2 years
AUC from time 0 to time dosing interval (AUCss,0-tau) | Approximately 2 years
CLss/Fss | Approximately 2 years
Vz/Fss | Approximately 2 years
accumulation ratio of Cmax (RCmax) after multiple doses | Approximately 2 years
accumulation ratio of AUC (RAUC) after multiple doses | Approximately 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Shanghai Jiao Tong University School of Medicine-Ruijin Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No